CLINICAL TRIAL: NCT02001779
Title: Study of Stent Insertion Combined With or Without Brachytherapy in Patients With Inoperable Malignant Biliary Obstruction
Brief Title: IRS(Irradiation Stent) vs. CS(Conventional Stent) Insertion in Inoperable Malignant Biliary Obstruction
Acronym: IRCSMBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Professor of Radiology & Chair,Department of Radiology, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR-C-STENT-MBO-83272121
Record Dates: First submitted 2013-11-22; First posted 2013-12-05 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Malignant Biliary Obstruction
Keywords: Malignant biliary obstruction; Obstruction/stricture; Stent; Brachytherapy; Bile duct
MeSH Terms: conditions — Bites and Stings; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biliary SEMS loaded with 125I seeds (Experimental): A self-expandable metallic biliary stent loaded with 125 iodine seeds is inserted in patients with inoperable malignant biliary obstruction.
  Interventions: Device: Biliary SEMS loaded with 125I seeds
- Conventional biliary SEMS (Active Comparator): A self-expandable metallic biliary stent is inserted in patients with inoperable malignant biliary obstruction.
  Interventions: Device: Conventional biliary SEMS

INTERVENTIONS:
Device: Biliary SEMS loaded with 125I seeds — A self-expandable metallic biliary stent loaded with 125 iodine seeds is inserted in patients with inoperable malignant biliary obstruction.
  Arms: Biliary SEMS loaded with 125I seeds
Device: Conventional biliary SEMS — A self-expandable metallic stent is inserted in patients with inoperable malignant biliary obstruction.
  Arms: Conventional biliary SEMS

SUMMARY:
Stenting the malignant biliary obstruction is considered to be the preferred palliation modality to relieve pruritus,cholangitis,pain and jaundice in patients without surgical indications of malignant biliary obstruction.An unicentral clinical trial has demonstrated the safety and technical feasibility of an irradiation biliary stent insertion in patients with biliary obstruction caused by adenocarcinomas, such a treatment seems have benefits in relieving jaundice and extending survival when compared to a conventional biliary stent.However,the small sample size,the population distribution of two groups will influence the final results in obtaining a powerful statistical conclusion.Therefore,a multicentric study was designed to prospectively compared the responses to the treatment with this irradiation biliary stent versus the conventional biliary self-expandable stent in patients with inoperable malignant biliary obstruction.

DETAILED DESCRIPTION:
Malignant biliary obstruction is a common condition caused by various carcinomas.The clinical process is usually silent and insidious,only 10-20% patients can be surgically removed once obstructive jaundice occurred.The long-term survival rate after resection remain dismal.Relief of obstructive jaundice plays major role on prognosis in patients without surgical indications.For unresectable patients,stenting the biliary obstruction is considered to be the preferred palliation modality to relieve pruritus,cholangitis,pain and jaundice.Although a number of new techniques for treatment of malignant biliary obstruction have been developed,there have been no significant differences in survival or quality of life comparing surgery bypass versus plastic stent insertion,metal stent insertion versus plastic stents insertion,or covered stent versus uncovered stents insertion in such patients.Our previous unicentric clinical trial has demonstrated the safety and technical feasibility of a biliary intraluminal irradiation stent insertion in patients with biliary obstruction caused by adenocarcinomas, such a treatment seems have benefits in relieving jaundice and extending survival when compared to a conventional biliary stent.However,the small sample size,the population distribution of two groups will influence the final results in obtaining a powerful statistical conclusion in the overall survival and stent patency between two groups.Therefore,a multicentric study was designed to prospectively compared the responses to the treatment with this irradiation biliary stent versus the conventional biliary self-expandable stent in patients with inoperable malignant biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Clinical,histological or pathological diagnosis of malignant biliary obstruction
* Unresectability or refusal to be surgically treated
* The Eastern Cooperative Oncology Group(ECOG) scores from 0 to 3
* With symptoms such as jaundice related to biliary obstruction
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Biliary obstruction of Bismuthe-Corlette,type I and II

Exclusion Criteria:

* Benign biliary obstruction
* The Eastern Cooperative Oncology Group(ECOG) score of 4
* Biliary tract stricture that could not be dilated enough to pass the delivery system
* Presence of metallic biliary stent or bile duct surgery
* Percutaneous transhepatic cholangiography(PTC) procedure was contraindicated
* Active hepatitis
* Biliary obstruction of Bismuthe-Corlette,type Ⅲ and Ⅳ
* Uncooperative or could not provide authorization and signature

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Patency | Participants will be followed till die or lost to follow-up,an expected average of a year.
  Time from stenting to the day when stricture/obstruction of the stent occured or restricture/reobstruction after recanalization the obstructed stent.

SECONDARY OUTCOMES:
Over survival | Participants will be followed till die or lost to follow-up,an expected average of a year.
  Time from stenting to the day when the patients died or lost to the follow-up.
Clinical success | Participants will be followed till die or lost to follow-up,an expected average of a year.
  The rate of relief of the symptoms and signs of the patients.
Safety | Participants will be followed till die or lost to follow-up,an expected average of a year.
  Including technique success rate,side effect/complication,radioactive safety.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, Ph.D,MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu HD, Guo JH, Huang M, Ji JS, Xu H, Lu J, Li HL, Wang WH, Li YL, Ni CF, Shi HB, Xiao EH, Lv WF, Sun JH, Xu K, Han GH, Du LA, Ren WX, Li MQ, Mao AW, Xiang H, Zhang KX, Min J, Zhu GY, Su C, Chen L, Teng GJ. Irradiation stents vs. conventional metal stents for unresectable malignant biliary obstruction: A multicenter trial. J Hepatol. 2018 May;68(5):970-977. doi: 10.1016/j.jhep.2017.12.028. Epub 2018 Jan 10. PMID 29331343